CLINICAL TRIAL: NCT06558266
Title: Comparison of Mental Imagery Ability According to Menstrual Cycle Phases
Brief Title: Mental Imagery in Menstrual Cycle Phases
Status: Completed | Type: Observational
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Asst. Prof., Izmir University of Economics
Other Study IDs: B.30.2.İEÜSB.0.05.05-20-291
Record Dates: First submitted 2024-07-29; First posted 2024-08-16 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-08

CONDITIONS: Menstruation; Mental Imagery; Menstrual Cycles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- menstrual cycle monitoring group: Female students between 18-25 with regular menstrual cycles
  Interventions: Other: Since this was an observational study, no intervention was performed.

INTERVENTIONS:
Other: Since this was an observational study, no intervention was performed. — Since it is an observational study, only evaluation will be made. Each participant s mental imagery ability will be evaluated with the Movement Imagery Vividness Questionnaire-2 four times, follicular phase, ovulation, luteal phase and menstrual phase. In addition, the pain intensity experienced during menstruation will be evaluated with the Numerical Classification Scale-11, and the symptoms experienced due to menstruation will be evaluated with the Menstruation Symptom Scale.

SUMMARY:
Hormonal fluctuations occur during the menstrual cycle and can affect cognition. For example, an increase in estrogen levels has been reported to temporarily enhance auditory perception of newly formed stimuli. It has been suggested that fluctuations in hormone levels can alter cognitive performance throughout the menstrual cycle because these fluctuations impact the neurobiology of the brain regions involved in cognition and emotion processing. Mental imagery (MI) refers to the mental process in which an individual imagines performing a movement without actually executing the movement. The effects of hormonal fluctuations on cognitive-perceptual skills have been mentioned above. In light of the above information, this study was planned to examine the relationship between menstrual symptom characteristics and mental imagery ability and to compare women s mental imagery abilities according to the phases of the menstrual cycle.

ELIGIBILITY:
Inclusion criteria

* Being a woman between the ages of 18-25,
* Having a regular menstrual cycle,
* Being a volunteer Exclusion criteria
* Using neuropsychiatric medication that may affect perception and cognitive skills.

People who do not participate in any of the four assessments will be excluded from the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The universe of the study consists of female students studying at Izmir University of Economics. With the permission of the Dean of the Faculty of Health Sciences of Izmir University of Economics, an announcement e-mail will be sent to all female students to inform them about the study and a list of volunteers will be created via the participation link. 151 female students who meet the study criteria will be included with the systematic sampling method. An "Informed Volunteer Consent Form" will be obtained from individuals who accept to participate in the study.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Motor Imagery Skill | In 1 month period
  The Vividness of Movement Imagery Questionnaire-2 will be used to assess the vividness of participants' movement imagery ability. In the questionnaire, a total of 12 different actions are imagined, and the questionnaire has three subscales (Internal Visual Imagery, External Visual Imagery, and Kinesthetic Imagery). A 5-point Likert scale (1: Perfectly clear and vivid as a normal vision - 5: No image at all: Only know you are thinking of the movement) is used to score each action, and the total score for each subscale ranges from 1 to 60.

SECONDARY OUTCOMES:
Menstrual Symptoms | at baseline
  The Menstruation Symptom Scale is one of the scales that evaluates the symptoms experienced due to menstruation in detail. It is a five-point Likert-type scale consisting of twenty-four items. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The MSÖ score is calculated by taking the total score average of the items in the scale. An increase in the score average indicates an increase in the severity of menstrual symptoms. The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints', 'Menstrual Pain' and 'Abdominal Pain'. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions.
Menstrual Pain | at baseline
  The numbered classification scale-11 (NSS-11) (0-10) will be used to evaluate menstrual pain. It is a practical and simple method recommended to evaluate the severity and variations of menstrual pain. The participant will be asked to give a score between 0-10 for the severity of pain they perceive/feel during menstruation. "0 means no complaints", "10 means very severe complaints"

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yakıt Yeşilyurt, PhD, Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No